CLINICAL TRIAL: NCT00383929
Title: A Double Blind, Randomised, 3-Arm Parallel Group, Multicentre, 8-Week, Phase III Study to Assess Antihypertensive Efficacy and Safety of the Combination of Candesartan Cilexetil (CC) /HCT 32/12.5mg and 32/25mg vs. CC 32mg Alone in Patients With Inadequate BP Control on Monotherapy With CC 32mg
Brief Title: Antihypertensive Efficacy and Safety of Candesartan/HCT 32/12.5 and 32/25 mg in Comparison With Candesartan 32 mg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2456C00001; Eudract No. 2005-005718-19
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Hypertension
Keywords: Blood pressure reduction; combination therapy; candesartan cilexetil; hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Candesartan Cilexetil (CC) /HCT 32/12.5mg
  Interventions: Drug: Candesartan cilexetil; Drug: Hydrochlorothiazide
- 2 (Experimental): Candesartan Cilexetil (CC) /HCT 32/25mg
  Interventions: Drug: Candesartan cilexetil; Drug: Hydrochlorothiazide
- 3 (Experimental): Candesartan Cilexetil monotherapy
  Interventions: Drug: Candesartan cilexetil

INTERVENTIONS:
Drug: Candesartan cilexetil — 32mg oral
  Other Names: ATACAND
Drug: Hydrochlorothiazide — 12.5 mg oral
  Other Names: HCTZ
  Arms: 1
Drug: Hydrochlorothiazide — 25 mg oral
  Other Names: HCTZ
  Arms: 2

SUMMARY:
In this study it is intended to compare the blood pressure lowering effect of the combination of candesartan cilexetil (candesartan) 32 mg and hydrochlorothiazide (HCT) 25 mg and the combination of candesartan 32 mg and HCT 12.5 mg to that of candesartan 32 mg alone in patients whose blood pressure is not well controlled on candesartan 32 mg monotherapy. The Primary Objectives are to compare sitting BP lowering effect of candesartan/HCT 32/25 mg and candesartan/HCT 32/12.5 mg with that of candesartan 32 mg, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for enrolment into the study (Visit 1) if they fulfil all of the following criteria:
* Provision of signed Informed Consent
* Primary hypertension, untreated or treated with a maximum of 2 antihypertensive drugs, which the patient and the physician are willing to withdraw at enrolment and change to candesartan monotherapy
* Mean sitting DBP 90-114 mmHg
* Patients will be eligible for randomisation (Visit 4) if they fulfil the following criterion:
* Mean sitting DBP 90-114 mmHg on treatment with candesartan 32 mg monotherapy (after 2 weeks with candesartan 16 mg and 6 weeks with candesartan 32 mg monotherapy). The run-in period should not be shorter than 8 weeks.

Exclusion Criteria:

* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff, CRO staff or staff at the investigational centre)
* Pregnant or lactating women, or women of childbearing potential not practising an adequate method of contraception eg, intrauterine device, oral contraception or progesterone implant and verified by a negative pregnancy test at Visit 1
* Secondary or malignant hypertension
* Sitting SBP of 180 mmHg or more
* Patients who are treated with candesartan 16 mg in combination with a diuretic or with candesartan 32 mg with or without any additional antihypertensive treatment
* Myocardial infarction, stroke, coronary bypass surgery or transient ischaemic attack within 6 months before enrolment
* Angina pectoris requiring more treatment than short-acting nitrates
* Chronic use of NSAIDs
* Aortic or mitral valve stenosis
* Cardiac failure requiring treatment
* Cardiac arrhythmia requiring treatment
* Gout
* Renal artery stenosis or kidney transplantation
* Intravascular volume depletion
* Hypersensitivity to any component of the investigational products
* Concomitant disease which may interfere with the assessment of the patient
* Past or present alcohol or drug abuse, or any condition associated with poor compliance
* Chronic liver disease or known liver enzyme values above three times the upper limit of the reference range for S-ASAT or S-ALAT
* Concomitant or previous treatment with other investigational drugs within 20 days of enrolment
* Previous enrolment in the present study
* S-creatinine of 180 μmol/l or above for men and of 140 μmol/l or above for women
* S-sodium or S-potassium outside the reference range
* Less than 85% compliance with study medication during the run-in phase

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1979 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Change (reduction) in sitting BP (24 hours after dose) | Assessed from baseline (randomisation) to the end of the study.

SECONDARY OUTCOMES:
Proportion of patients with controlled sitting BP in each treatment group | Assessed at the end of the study
Occurrence of Adverse Events and discontinuation of study medication due to AEs from baseline (randomisation) to the end of the study | Assessed from baseline (randomisation) to the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Established Brands HTN/CHF Medical Sience Director, MD, Study Director — AstraZeneca; Gerd Bonner, MD, Principal Investigator — MEDIAN Kliniken Bad Krozingen
Locations (132):
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Copenhagen
  - Research Site, Frederiksberg
  - Research Site, Herlev
  - Research Site, Vejle
- Estonia (4):
  - Research Site, Pärnu
  - Research Site, Tallinn
  - Research Site, Tartu
  - Research Site, Võru
- France (14):
  - Research Site, Albens
  - Research Site, Arras
  - Research Site, Béziers
  - Research Site, Broglie
  - Research Site, Chartres
  - Research Site, Gémenos
  - Research Site, Hinx
  - Research Site, Husseren-Wesserling
  - Research Site, Labarthe-sur-Lèze
  - Research Site, Rosiers-d'Égletons
  - Research Site, Seraincourt
  - Research Site, Strasbourg
  - Research Site, Tours
  - Research Site, Vourey
- Germany (33):
  - Research Site, Augsburg
  - Research Site, Bad Krozingen
  - Research Site, Bad Segeberg
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Cloppenburg
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Goch
  - Research Site, Großheirath
  - Research Site, Hamburg
  - Research SIte, Hann
  - Research Site, Hermaringen
  - Research Site, Herne
  - Research Site, Karlsruhe
  - Research Site, Kiel
  - Research Site, Kippenheim
  - Research Site, Künzing
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Nuremberg
  - Research Site, Riesa
  - Research Site, Rodgau-dudenhofen
  - Research Site, Schwerin
  - Research Site, Siegen
  - Research Site, Steinfurt
  - Research Site, Straßkirchen
  - Research Site, Tübingen
  - Research Site, Werne
  - Research Site, Witten
- Lithuania (5):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Panevezys
  - Research Site, Šiauliai
  - Research Site, Vilnius
- Netherlands (19):
  - Research Site, 's-Gravenzande
  - Research Site, 's-Hertogenbosch
  - Research Site, Bennebroek
  - Research Site, Deurne
  - Research Site, Echt
  - Research Site, Ermelo
  - Research Site, Hengelo
  - Research Site, Hoogvliet
  - Research Site, Lichtenvoorde
  - Research Site, Losser
  - Research Site, Musselkanaal
  - Research Site, Oude Pekela
  - Research Site, Rijswijk
  - Research Site, Roelofarendsveen
  - Research Site, Rotterdam
  - Research Site, The Hague
  - Research Site, Volendam
  - Research Site, Woerden
  - Research Site, Zaandam
- Poland (11):
  - Research Site, Chrzanów
  - Research Site, Elblag
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Oława
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Skierniewice
  - Research Site, Szczecin
- Serbia and Montenegro (5):
  - Research Site, Belgrade
  - Research Site, Niska Banja
  - Research Site, Nis
  - Research Site, Sremska Kamenica
  - Research Site, Zemun
- Sweden (9):
  - Research Site, Boden
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Linköping
  - Research Site, Malmo
  - Research Site, Motala
  - Research Site, Örebro
  - Research Site, Skellefteå
  - Research Site, Uppsala
- Ukraine (6):
  - Research Site, Chenoutsy
  - Research Site, Dnipro
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
- United Kingdom (20):
  - Research Site, Addlestone
  - Research Site, Ashford
  - Research Site, Ayrshire
  - Research Site, Burbage
  - Research Site, Cheadle
  - Research Site, Chesterfield
  - Research Site, Coventry
  - Research Site, Ely
  - Research Site, FIFE
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Hastings
  - Research Site, Helensburgh
  - Research Site, Morriston
  - Research Site, Motherwell
  - Research Site, Newton Mearns
  - Research Site, Northwood Middlesex
  - Research Site, Paignton
  - Research Site, Royal Leamington Spa
  - Research Site, Wokingham